CLINICAL TRIAL: NCT00628017
Title: The Effects of Omega-3 Fatty Acids Monotherapy in Alzheimer's Disease and Mild Cognitive Impairment: a Preliminary Randomized Double-Blind Placebo-Controlled Study
Brief Title: Preliminary Study of Fish Oil and Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Psychiatric Center, Taiwan (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Chih-Chiang Chiu, M.D., Department of Psychiatry, Taipei City Psychiatric Center, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOH-92-TD-1095
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: polyunsaturated fatty acids; Alzheimer's disease; mild cognitive impairment; fish oil; cognition
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): omega-3 PUFAs(180mg eicosapentaenoic acid[EPA] + 120mg docosahexaenoic acid[DHA]/capsule), 3 capsules twice daily, total daily omega-3 fatty acid dosage of 1080 mg of EPA and 720 mg of DHA
  Interventions: Dietary Supplement: omega-3 polyunsaturated fatty acids ( EPA+DHA)
- 2 (Placebo Comparator): three identical placebo capsules twice daily which contained olive oil esters.
  Interventions: Dietary Supplement: omega-3 polyunsaturated fatty acids ( EPA+DHA)

INTERVENTIONS:
Dietary Supplement: omega-3 polyunsaturated fatty acids ( EPA+DHA) — Group 1 received omega-3 PUFAs as 3 capsules twice daily (total daily omega-3 fatty acid dosage of 1080 mg of EPA and 720 mg of DHA). Group 2 received three identical placebo capsules twice daily which contained olive oil esters. Identical gelatin capsules were used. Both treatment and placebo capsules were vacuum deodorized and supplemented with tertiary-butyl hydroquinone, 0.2 mg/g, and tocopherols, 2 mg/g, as antioxidants. The source of the omega-3 fatty acids was menhaden fish body oil concentrate.
  Other Names: fish oil; n3 fatty acids

SUMMARY:
This preliminary study is aimed to investigate whether it is feasible to conduct a study to use fish oil compared to the placebo(olive oil) in people with cognitive impairment. We will also explore whether fish oil has better efficacy in some clinical aspects in people with cognitive impairment during 24 weeks intervention. The major clinical outcome will be:

1. general clinical impression
2. cognitive function

DETAILED DESCRIPTION:
Despite some positive findings from observational and animal studies, the effects of n-3 PUFA administration on cognitive impairment in humans have received little evaluation to date. Although some clinical trials of fish oil have been reported, the results are inconsistent. Given these inconsistent findings, we carried out a preliminary study to investigate the effect of fish oil monotherapy on cognitive function and general clinical condition in patients with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled the diagnosis of AD according to the American Psychiatric Association, DSM-IV criteria, with mild or moderate severity( defined by an Mini Mental Status Examination (MMSE) score between 10 and 26, and a Clinical Dementia Rating (CDR) score of 1 or 2.)
* or amnesic MCI( defined as (1). Subjective memory impairment by the patient and /or an informant, (2) objective memory impairment falling at least 1.5 standard deviations or more below age- and education-specific norms on the Logical Memory delayed-recall score from the Wechsler Memory Scale III (3) relatively normal performance in other cognitive domains, (4) no impairment in activities of daily living, and (5) failure to meet DSM-IV criteria for dementia.)

Exclusion Criteria:

* inadequate motor or sensory capacity to comply with testing
* any ischemic lesion on brain CT reported by the radiologist or a modified Hachinski Ischemic Scale score >4
* a 17-item Hamilton Depression Scale (HDRS)score > 13
* abnormal levels of folic acid, vitamin B12, or thyroid function
* severe comorbidity, including another neurodegenerative diseases, another chronic debilitating neurological illness (e.g. cerebral palsy), brain trauma, tumors, severe pulmonary, renal, liver disease, cardiac disease, or autoimmune disease, or conditions expected to cause death within one year.
* Participants with a diagnosis of alcoholism, schizophrenia, and bipolar disorder were excluded.
* Participants receiving cholinesterase agents during the screen or taking NSAID on a long-term basis

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-01; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
the Clinician's Interview-Based Impression of Change Scale (CIBIC-plus) | 24 weeks
the cognitive portion of the Alzheimer's Disease Assessment Scale (ADAS-cog) | 24 weeks

SECONDARY OUTCOMES:
Mini Mental Status Examination (MMSE) scores | 24 weeks
17-item Hamilton Depression Scale (HDRS) | 24 weeks
adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chiang Chiu, M.D., Principal Investigator — Department of Psychiatry, Taipei Psychiatric Center, Taipei City Hospital, Taipei, Taiwan; Shih-Yi Huang, PhD., Principal Investigator — School of Nutrition and Health Sciences, Taipei Medical University, Taiwan
Locations (1):
- Taipei City Psychiatric Center, Taipei City Hospital, Taipei, Taiwan